CLINICAL TRIAL: NCT01846195
Title: Clinical Evaluation of the Zynex Blood Volume Monitor (CM-1500) in Healthy Adult Patients During a Blood Draw
Brief Title: Evaluation of the Zynex Blood Volume Monitor in Healthy Adult Patients During a Blood Draw
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zynex Monitoring Solutions (Industry)
Collaborators: DTarget (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Zynex500
Record Dates: First submitted 2013-03-13; First posted 2013-05-03 (Estimated); Results first posted 2022-11-09 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-10

CONDITIONS: Blood Loss
Keywords: blood loss
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- no blood draw (Sham Comparator): CM 1500 with no blood draw
  Interventions: Device: CM 1500
- blood draw (Active Comparator): CM 1500 with blood draw
  Interventions: Device: CM 1500

INTERVENTIONS:
Device: CM 1500

SUMMARY:
Non-invasive monitoring to measure changes in blood volume.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Between 18-35 years of age
* Weight between 130-200 pounds

Exclusion Criteria:

* Known cardiac disease
* Recent caffeine intake
* Tobacco use in the (4) hours prior to screening
* Infection
* Pregnancy
* Hemoglobin <13.5 g/dl

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2012-06-06 (Actual); Primary Completion 2013-03-20 (Actual); Study Completion 2013-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Ziegler, MD, Principal Investigator — Premier Research
Locations (1):
- Premier Research Group, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- no Blood Draw: CM 1500 with no blood draw
  CM 1500
- Blood Draw: CM 1500 with blood draw
  CM 1500
Period: Overall Study
Arm/Group | no Blood Draw | Blood Draw
Started | 5 | 45
Completed | 5 | 45
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | no Blood Draw | Blood Draw | Total
Number analyzed (Participants) | 5 | 45 | 50
Age, Continuous [Median (Full Range); unit: years] | 25.5 [18 to 33] | 25.9 [18 to 34] | 25.7 [18 to 34]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 21 | 23
  Male | 3 | 24 | 27
Region of Enrollment [Number; unit: participants]
  United States | 5 | 45 | 50
Height [Mean (Full Range); unit: inches] | 69.2 [65 to 73] | 67.9 [62 to 75] | 68.6 [62 to 75]
Weight [Mean (Full Range); unit: pounds] | 162.3 [136 to 196] | 158.4 [134 to 196] | 160.4 [134 to 196]

OUTCOME MEASURES:

1. Primary Outcome: Detect by Non-invasive Monitoring a Change in Blood Volume During a Whole Blood Draw
Description: Detection by non-invasive monitoring a change in blood volume (yes or no) during a whole blood draw
Time Frame: At study completion (completion of blood draw)
Population: Number of subjects for which blood loss was detected.
Measure: Number; unit: participants
Arm/Group | no Blood Draw | Blood Draw
Number analyzed (Participants) | 5 | 45
participants | 0 | 45

ADVERSE EVENTS:
Time Frame: Adverse event data was collected through the completion of the study. Adverse events per subject may have occurred during the blood draw or within 24 hours following with any potential reaction to electrode adhesive.
Arm/Group | no Blood Draw | Blood Draw
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/45
Other Adverse Events (participants affected / at risk) | 0/5 | 5/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | no Blood Draw (N=5) | Blood Draw (N=45)
Vasovagal Reaction to Blood Draw (General disorders) | 0 | 5 — Several subjects had a vasovagal reaction to the blood draw. Specifically, subject reported being lightheaded or dizzy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No